CLINICAL TRIAL: NCT05612204
Title: Evaluation of Targeted Prostate Biopsies Under MRI: Tolerance and Contribution in the Therapeutic Decision - Exploratory Study
Acronym: BIOPROSTATIRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A00792-41
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy under MRI (Experimental)
  Interventions: Procedure: Biopsy under MRI

INTERVENTIONS:
Procedure: Biopsy under MRI — Biopsy under MRI

SUMMARY:
The goal of this clinical trial is to assess the concordance of treatment decisions made in multidisciplinary consultation meeting based on targeted biopsies alone or targeted biopsies associated with systematic biopsies in patients with suspected prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer in France and is the third most common cancer death in men.

Early detection is based on family and ethnic history, digital rectal examination and total PSA testing. It is done at age 50 for the general population but is restricted to men with an estimated survival of more than 10 years.

In case of clinical suspicion of prostate cancer, the diagnosis is based on the realization of prostate biopsies. Until recently, 12 so-called "systematic" (BS) biopsies were performed under ultrasound control, according to a standardized protocol, which allowed sampling of the entire prostate.

Since the latest recommendations of the French Association of Urology in 2020, an MRI is systematically indicated before performing biopsies. Indeed, MRI is a sensitive technique that will increase the suspicion of significant prostate cancer. An MRI is considered "positive" if at least one suspicious area with a PI-RADS score ≥ 3 is detected. In this case, the French Association of Urology recommends performing so-called targeted biopsies (BC) on these suspicious areas associated with the 12 SBs.

From a technical point of view, ultrasound is the reference examination for performing targeted biopsies on suspicious lesions detected on MRI, either by visual guidance (cognitive identification) or by image fusion techniques, MRI and ultrasound.

It is now technically possible to perform biopsies directly under MRI in clinical practice, but the development of this approach remains limited in France. This technique makes it possible to biopsy the suspect area without resorting to image fusion, thus limiting targeting errors.

As only MRI can detect cancerous lesions, this study is based on the hypothesis that targeted biopsies alone taken under MRI could make it possible to make a therapeutic decision within the framework of a multidisciplinary consultation meeting (RCP) without resorting to systematic biopsies under ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male, aged between ≥ 50 and ≤ 75 years old
* Patient with no history of prostate biopsy
* Patient with a PSA greater than 4 and/or a pathological digital rectal examination
* Patient having an MRI of interpretable quality carried out within the HPA
* Patient with a single lesion with a PI-RADS score ≥ 3
* Affiliated patient or beneficiary of a social security scheme
* French-speaking patient who signed an informed consent

Exclusion Criteria:

* Patient with a contraindication to MRI
* Patient with multiple targets
* Patient with lesions with PI-RADS score 1 and 2
* Patient on long-term anticoagulants and unable to stop it
* Patient already included in another study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Patient hospitalized without consent

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Type of care offered in multidisciplinary consultation meeting | 2 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- HPA, Antony, France

IPD SHARING:
Plan to Share IPD: No